CLINICAL TRIAL: NCT02021006
Title: Antibiotic Prophylaxis and Renal Damage In Congenital Abnormalities of the Kidney and Urinary Tract
Acronym: PREDICT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Ministero della Salute, Italy (Other); IL Sogno di Stefano (Other)
Responsible Party: Principal Investigator, Giovanni Montini, Prof., Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREDICT trial
Record Dates: First submitted 2013-12-01; First posted 2013-12-27 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Vesicoureteral Reflux; Renal Hypodysplasia, Nonsyndromic, 1; Chronic Kidney Disease
Keywords: antibiotic prophylaxis; vesicoureteral reflux; congenital abnormalities of kidney; renal hypodysplasia; chronic kidney disease
MeSH Terms: conditions — Vesico-Ureteral Reflux; Renal Hypodysplasia, Nonsyndromic, 1; Renal Insufficiency, Chronic | interventions — Nitrofurantoin; Amoxicillin-Potassium Clavulanate Combination; Amoxicillin; Clavulanic Acid; Trimethoprim, Sulfamethoxazole Drug Combination; Cefixime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ANTIBIOTIC PROPHYLAXIS (Active Comparator): Children in this arm will take antibiotic prophylaxis for 2 years. Patients in this arm will do clinical/instrumental follow-up for 5 years.
  The antibiotic for prophylaxis will be chosen by Physicians according to the local resistance spectrum of bacteria responsible of UTIs
  Physicians can chose one the following schedules:
  * nitrofurantoin 1.5-2 mg/kg per day
  * Amoxicillin-Potassium Clavulanate Combination 15 mg/kg per day (dose expressed in units equivalent to amoxicilline)
  * cefixime 2 mg/kg per day
  * trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)
  Interventions: Drug: nitrofurantoin; Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Trimethoprim/sulfamethoxazole; Drug: Cefixime
- NO PROPHYLAXIS (Experimental): Children in this arm will not take antibiotic prophylaxis. Patients in this arm will do clinical/instrumental follow-up for 5 years
  Interventions: Other: No prophylaxis

INTERVENTIONS:
Drug: nitrofurantoin — antibiotic prophylaxis of urinary tract infections The antibiotic for prophylaxis will be chosen by Physicians according to the local resistance spectrum of bacteria responsible of UTIs
  Physicians can chose one the following schedules:
  * nitrofurantoin 1.5-2 mg/kg per day
  * amoxicilline/clavulanic acid 15 mg/kg per day (dose expressed in units equivalent to amoxicilline)
  * cefixime 2 mg/kg per day
  * trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)
  Other Names: Furadantin
  Arms: ANTIBIOTIC PROPHYLAXIS
Other: No prophylaxis — children will be followed, but no antibiotic prophylaxis will be administered
  Arms: NO PROPHYLAXIS
Drug: Amoxicillin-Potassium Clavulanate Combination — antibiotic prophylaxis of urinary tract infections The antibiotic for prophylaxis will be chosen by Physicians according to the local resistance spectrum of bacteria responsible of UTIs
  Physicians can chose one the following schedules:
  * nitrofurantoin 1.5-2 mg/kg per day
  * amoxicilline/clavulanic acid 15 mg/kg per day (dose expressed in units equivalent to amoxicilline)
  * cefixime 2 mg/kg per day
  * trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)
  Other Names: amoxicilline/clavulanic acid, augmentin, clavulin
  Arms: ANTIBIOTIC PROPHYLAXIS
Drug: Trimethoprim/sulfamethoxazole — antibiotic prophylaxis of urinary tract infections The antibiotic for prophylaxis will be chosen by Physicians according to the local resistance spectrum of bacteria responsible of UTIs
  Physicians can chose one the following schedules:
  * nitrofurantoin 1.5-2 mg/kg per day
  * amoxicilline/clavulanic acid 15 mg/kg per day (dose expressed in units equivalent to amoxicilline)
  * cefixime 2 mg/kg per day
  * trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)
  Other Names: bactrim
  Arms: ANTIBIOTIC PROPHYLAXIS
Drug: Cefixime — antibiotic prophylaxis of urinary tract infections The antibiotic for prophylaxis will be chosen by Physicians according to the local resistance spectrum of bacteria responsible of UTIs
  Physicians can chose one the following schedules:
  * nitrofurantoin 1.5-2 mg/kg per day
  * amoxicilline/clavulanic acid 15 mg/kg per day (dose expressed in units equivalent to amoxicilline)
  * cefixime 2 mg/kg per day
  * trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)
  Other Names: cefixoral
  Arms: ANTIBIOTIC PROPHYLAXIS

SUMMARY:
The exact role of urinary tract infection in the appearance of chronic kidney disease is unclear. Children with congenital malformations of kidney and urinary tract have the higher risk of impairment of renal function. To understand if the use of antibiotic prophylaxis can reduce the risk of urinary tract infection in children with these malformations, this study will randomize children in two groups. Group A will not take antibiotic prophylaxis, Group B will take antibiotic prophylaxis for 2 years. This study will assess if antibiotic prophylaxis reduce the risk of urinary tract infections in these children and if urinary tract infections influence the appearance of renal damage.

Our hypothesis is that prophylaxis reduce the risk of infection in severe vesicoureteral reflux and that urinary tract infections, in morphologically normal kidneys, will not result in chronic renal failure.

DETAILED DESCRIPTION:
Bacterial urinary tract infections (UTI) are common in young children. The presence of fever is considered to be a marker of renal parenchymal involvement. Renal damage during the acute phase of infection may lead to scarring, yet the role that scarring plays in the appearance of chronic kidney failure is unknown. It is also unclear what influence scars have on the natural course of kidney function, especially in children with renal hypodysplasia, with or without vesicoureteral reflux (VUR). Renal hypodysplasia is the most common cause for dialysis and transplantation in the pediatric population.

Patients suffering from recurrent UTIs and VUR have often undergone corrective surgery. For many years, it was also thought necessary to prescribe long-term antibiotic prophylaxis to all children with VUR. These treatment strategies were based on the ideas and opinions of the experts, rather than on hard scientific evidence. As regards the prevention of recurrent UTIs and the subsequent development of renal scarring, a long-term international study on Reflux was not able to demonstrate that surgical correction is more effective than antibiotic prophylaxis. Very little data is available regarding the use of long-term antibiotic prophylaxis in children with high grade reflux with or without renal hypodysplasia.

The use of antibiotics during the first few months of life has been associated with a significant increase in body mass index (BMI). Even though this effect is probably limited, it could have a significant impact on public health given the widespread use of antibiotics and due to the considerable increase in cases of pediatric and adult obesity seen over the last few years.

In spite of the lack of evidence, the use of prophylaxis is largely routine practice in most centres. Therefore, a randomized study is necessary in order to evaluate whether prophylaxis reduces the risk of symptomatic infections and subsequent renal damage.

To assess the role of prophylaxis in patient with high grade vesicoureteral reflux we will perform a multicentre, prospective, randomized, controlled, open-label, study.

Patients enrolled will be randomized in two groups:

Group A: no antibiotic prophylaxis. Group B: antibiotic prophylaxis for 24 months. The choice of which antibiotic to prescribe from the list below is left to the discretion of each investigator, on the basis of local antibiotic resistance patterns.

* nitrofurantoin 1.5-2 mg/kg per day
* amoxicilline/clavulanic acid 15 mg/kg per day (dose expressed in units equivalent to amoxicillin)
* cefixime 2 mg/kg per day
* trimethoprim/sulfamethoxazole 2.5 mg/kg per day (dose expressed in units equivalent to trimethoprim)

The study is comprised of:

* Phase 1: Pre-randomization - screening tests to determine eligibility for the trial.
* Phase 2: Active treatment - this phase follows randomization and foresees 24 months of antibiotic prophylaxis for Group B and clinical surveillance for Group A.
* Phase 3: Follow-up - a further 36 months of clinical, laboratory and instrumental evaluation of renal function and the progression of renal damage for a total follow-up period of 5 years

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 and 4 months (> 4 weeks and <20 weeks of post-natal age)
* Gestational age > 35 weeks
* Glomerular filtration rate (calculated according to Schwartz) > 15 ml/min/1.73 m2
* No previous symptomatic UTI
* Imaging Diagnostic work-up completed and presence of grade III to V vesicoureteral reflux
* Informed consent of parents

Exclusion Criteria:

* Age <1 and >4 months
* Gestational age < 35 weeks
* Glomerular filtration rate (calculated according to Schwartz) < 15 ml/min/1.73 m2 at three months of age
* Patients with neurogenic bladder, myelomeningocele, ureteropelvic junction and/or ureterovesical junction obstruction, or other malformations leading to potential voiding disturbances.
* Presence of urethral valves
* Patients with no or low grade reflux (grade I and II).
* Hypersensitivity to the all the utilized antimicrobial agent
* Children with serious clinical conditions which, according to the investigator, prevent them from being included in the study cohort.
* Use of experimental drugs in the month previous to the beginning of the study
* Children unable to follow the established protocol procedures or whose parents are unable to sign the informed consent.

Ages: 1 Month to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 292 (Actual)
Dates: Start 2013-12; Primary Completion 2020-01 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
urinary tract infections rate | during the first 24 months from enrolment
  Urinary tract infections will be strictly monitored in all enrolled patients (both group A and group B). The rate of urinary tract infections in the first 24 months from the enrolment will be compared between 2 groups

SECONDARY OUTCOMES:
febrile urinary tract infections | during the first 24 months from enrolment
  Febrile urinary tract infections will be strictly monitored in all enrolled patients (both group A and group B). The rate of febrile urinary tract infections in the first 24 months from the enrolment will be compared between 2 groups
renal scars | at 2 years and 5 years from enrolment
  the appearance of renal scars in a dimercaptosuccinic acid (DMSA) scan will be detected at 2 and 5 years from enrolment and compared between the 2 groups.
serum creatinine (renal function) | at the enrolment,1 year, 2 years, 3 years, 4 years, 5 years
  The renal function (serum creatinine) will be monitored for all enrolled patients to explore the appearance and progression of renal damage
hypertension | at 4, 8, 12, 18, 24, 36, 48, 60 months from enrolment
  the appearance of hypertension will be monitored at every visit in all enrolled children
proteinuria | at 4, 8, 12, 18, 24, 36, 48, 60 months from enrolment
  the appearance of proteinuria will be monitored at every visit in all enrolled children
body mass index | at 2 and 5 years from enrolment
  body mass index will be evaluated at 2 and 5 years of follow-up and it will be correlated to the use of antibiotic prophylaxis
serum cystatin C (renal function) | at the enrolment,1 year, 2 years, 3 years, 4 years, 5 years
  The renal function (serum cystatin-C) will be monitored for all enrolled patients to explore the appearance and progression of renal damage
modification in gut microbiota induced by continuous antibiotic exposure during the first months of life | at the enrollment, 4 months, 8 months, 12 months, 2 years, 3 years, 4 years, 5 years
  A stool sample will be collected, frozen and stored for gut microbiota and resistome profile analysis

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Montini, MD, Study Chair — Pediatric Nephrology, Dialysis and Transplant Unit, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milan; Franz Schaefer, Professor, Study Director — Center for Pediatrics and Adolescent Medicine Division of Pediatric Nephrology, Heidelberg, Germany; Otto Mehls, Professor, Principal Investigator — Center for Pediatrics and Adolescent Medicine Division of Pediatric Nephrology, Heidelberg, Germany; Lutz T. Weber, Professor, Principal Investigator — Ärztlicher Leiter der Kindernephrologie Klinik und Poliklinik für Kinder- und Jugendmedizin Uniklinik Köln - Köln; Aleksandra M Zurowska, Professor, Principal Investigator — Medical University of Gdansk, Department Paediatric & Adolescent Nephrology & Hypertension - Gdansk - Poland; Fatos Yalcinkaya, Professor, Principal Investigator — Department of Pediatric Nephrology, School of Medicine, Ankara University, Ankara, Turkey; Esra Baskin, Professor, Principal Investigator — Paediatric Nephrology Division, Department of Paediatrics, Faculty of Medicine, Baskent University, Ankara, Turkey; Enrico Verrina, MD, Principal Investigator — UOC Nefrologia, Dialisi e Trapianto, IRCCS Giannina Gaslini, Genova, Italy; William Morello, MD, Principal Investigator — Pediatric Nephrology, Dialysis and Transplant Unit, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Milan; Piotr Czarniak, MD, Principal Investigator — Department of Nephrology, Transplantology and Internal Medicine, Medical University of Gdansk, Gdansk - Poland
Locations (1):
- Pediatric Nephrology Dialysis and Transplant Unit IRCCS Ca'Granda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morello W, Baskin E, Jankauskiene A, Yalcinkaya F, Zurowska A, Puccio G, Serafinelli J, La Manna A, Krzemien G, Pennesi M, La Scola C, Becherucci F, Brugnara M, Yuksel S, Mekahli D, Chimenz R, De Palma D, Zucchetta P, Vajauskas D, Drozdz D, Szczepanska M, Caliskan S, Lombet J, Minoli DG, Guarino S, Gulleroglu K, Ruzgiene D, Szmigielska A, Barbi E, Ozcakar ZB, Kranz A, Pasini A, Materassi M, De Rechter S, Ariceta G, Weber LT, Marzuillo P, Alberici I, Taranta-Janusz K, Caldas Afonso A, Tkaczyk M, Catala M, Cabrera Sevilla JE, Mehls O, Schaefer F, Montini G; PREDICT Study Group. Antibiotic Prophylaxis in Infants with Grade III, IV, or V Vesicoureteral Reflux. N Engl J Med. 2023 Sep 14;389(11):987-997. doi: 10.1056/NEJMoa2300161. Epub 2023 Sep 12. PMID 37702442